CLINICAL TRIAL: NCT06585358
Title: DoseTB-individualised Dosing by Model-informed Precision Dosing for Pulmonary Tuberculosis
Acronym: DoseTB
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Region Östergötland (Other)
Responsible Party: Principal Investigator, Lina Davies Forsman, Principal Investigator, Karolinska Institutet
Other Study IDs: 4-1624/2023
Record Dates: First submitted 2024-06-13; First posted 2024-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pulmonary
Keywords: model-informed precision dosing; individualised dosing
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary tuberculosis
  Interventions: Other: MIPD

INTERVENTIONS:
Other: MIPD — This is a non-inverventional study

SUMMARY:
The goal of this observational study is to investigate whether model-informed precision dosing (MIPD), as a clinical support for early individualised dosing in addition to the national TB care program, can optimise the drug exposure of TB drugs during TB treatment.

Main research questions:

In adult patients with drug-susceptible pulmonary tuberculosis, can current dose recommendations and information received from MIPD help clinicians in a timely manner to optimise the drug exposure of TB drugs in the early treatment phase, i.e., the time from PK sampling to dose adjustment (keep or adjust dose)?

Specific aims

I. To perform a process evaluation of early MIPD for rifampicin, isoniazid, pyrazinamide and ethambutol during active TB treatment.

II. To study the target attainment of first-line TB drugs with MIPD.

III. To evaluate model precision of predicted versus detected drug concentrations.

Drug concentrations will be measured in study participants during TB treatment, and drug exposure and the optimal dose will be predicted by MIPD using pharmacokinetic population models.

DETAILED DESCRIPTION:
Background:

Individualised treatment for tuberculosis (TB) to improve treatment outcome has still some substantial obstacles to pass before becoming a reality in clinical practice. Previous studies, including studies from the study research group, have shown that lower than recommended drug concentrations of TB drugs are common, and affect treatment outcome. Despite this, lower than recommended doses are often prescribed by clinicians. Adequate drug doses should be ensured as early as possible in the intensive phase when the bacterial load is high. Simple therapeutic drug monitoring (TDM) at the time of steady state of TB drugs are used in many clinical settings today, but time to dose adjustments to avoid suboptimal drug levels is typically several weeks. However, pharmacokinetic models are in place to guide individualised drug dosing by Model-Informed Precision Dosing (MIPD) already from the first days of treatment. MIPD, in combination with currently recommended dose recommendations, can be used to derive the most efficacious and safe dose for a patient. A similar approach has been implemented for dosing of vancomycin in children but has not been used in a clinical setting in the field of TB. This study will evaluate the logistics and dose regimens when clinicians are given the current dose recommendations of the first-line drugs rifampicin, isoniazid and pyrazinamide, as well as the results of the MIPD, for patients with active pulmonary TB.

ELIGIBILITY:
Inclusion criteria

1. Adult persons ≥18 years with confirmed pulmonary TB (established through Mtb cultures or PCR for Mtb by clinical routine)
2. Ongoing or planned treatment of TB that includes rifampin
3. Written informed consent

Exclusion criteria

1. TB treatment with rifampin for longer than 8 weeks prior to inclusion
2. TB treatment with intravenous rifampin (including patients treated at an intensive care unit (ICU) or patients with cerebral TB)
3. TDM of rifampin has already been performed (>24 h before inclusion) by clinical routine
4. Study participants with extrapulmonary TB without pulmonary TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion of study participants will be done prospectively at two hospitals included in the study sites (Karolinska University Hospital and Region Östergötland). Only patients with pulmonary TB will be included as the MIPD models have been developed using data sets of pulmonary TB and not for extrapulmonary TB.
  Participants who are unable to give an informed consent (e.g. persons with severe dementia) will not be included.
  The investigators will include at least 30 participants. Blood samples for drug concentration analysis will be performed 2+4 hours postdose at 2 -3 occasions during the study period and measure by a validated HPLC method at Clinical Pharmacology Laboratories in the regions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of predicted dose | Within the first 5 days from sampling
  Proportion of participants with predicted doses of rifampicin, isoniazid and/or pyrazinamide within 5 days from sampling (%)

SECONDARY OUTCOMES:
Proportion reaching predicted drug exposure | Through study completion, an average of one month
  For participants with dose-predicted treatment, proportion who will reach the target levels for rifampicin, isoniazid and/or pyrazinamide after MIPD
Model precision | Through study completion, an average of one month
  Precision of the model comparing predicted drug levels to the detected drug levels (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lina Davies Forsman, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulla A, Edwina EE, Flint RB, Allegaert K, Wildschut ED, Koch BCP, de Hoog M. Model-Informed Precision Dosing of Antibiotics in Pediatric Patients: A Narrative Review. Front Pediatr. 2021 Feb 23;9:624639. doi: 10.3389/fped.2021.624639. eCollection 2021. PMID 33708753
- [Background] Azuma J, Ohno M, Kubota R, Yokota S, Nagai T, Tsuyuguchi K, Okuda Y, Takashima T, Kamimura S, Fujio Y, Kawase I; Pharmacogenetics-based tuberculosis therapy research group. NAT2 genotype guided regimen reduces isoniazid-induced liver injury and early treatment failure in the 6-month four-drug standard treatment of tuberculosis: a randomized controlled trial for pharmacogenetics-based therapy. Eur J Clin Pharmacol. 2013 May;69(5):1091-101. doi: 10.1007/s00228-012-1429-9. Epub 2012 Nov 14. PMID 23150149
- [Background] Pasipanodya JG, McIlleron H, Burger A, Wash PA, Smith P, Gumbo T. Serum drug concentrations predictive of pulmonary tuberculosis outcomes. J Infect Dis. 2013 Nov 1;208(9):1464-73. doi: 10.1093/infdis/jit352. Epub 2013 Jul 29. PMID 23901086
- [Background] Niward K, Davies Forsman L, Bruchfeld J, Chryssanthou E, Carlstrom O, Alomari T, Carlsson B, Pohanka A, Mansjo M, Jonsson Nordvall M, Johansson AG, Eliasson E, Werngren J, Paues J, Simonsson USH, Schon T. Distribution of plasma concentrations of first-line anti-TB drugs and individual MICs: a prospective cohort study in a low endemic setting. J Antimicrob Chemother. 2018 Oct 1;73(10):2838-2845. doi: 10.1093/jac/dky268. PMID 30124844